CLINICAL TRIAL: NCT02269098
Title: The Synergy to Control Emergency Department Hyperglycemia Program for Type 2 Diabetes: STEP-Diabetes.
Brief Title: The Synergy to Control Emergency Department Hyperglycemia Program for Type 2 Diabetes
Acronym: STEP-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: American Diabetes Association (Other); Sanofi (Industry); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011-010
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2; Medication Adherence; HYPERGLYCEMIA
Keywords: type 2 diabetes; hyperglycemia; Emergency Department; Patient Education as Topic; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Medication Adherence; Hyperglycemia; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Diabetes survival skills self-management education; plus diabetes medication management using medication algorithm by diabetes educator supervised by endocrinologist, plus health system naviagation.
  Metformin, sulfonylureas and basal insulin were included in the algorithm. Survival skills DSME included: BG meter instruction if the patient did not already have a meter or confirmation of self-BG monitoring technique if they did; instructions on how to self-inject insulin if prescribed; and information on BG targets, signs and treatment of hypoglycemia and hyperglycemia, basic nutrition information and when to call the doctor or go to the ED.
  Interventions: Other: Diabetes medication management
- Control (No Intervention): Usual ED care was provided to controls. Hyperglycemia was treated with rapid acting insulin and with IV hydration, if indicated. DM medications were added and/or doses were adjusted at the discretion of the ED physician and prescriptions provided. Insulin, however, was not prescribed as a new medication due to staff concerns regarding post-discharge hypoglycemia and lack of certainty of timely medical follow-up. Follow-up with primary care was recommended.

INTERVENTIONS:
Other: Diabetes medication management — As above plus- Follow-up intervention visits were at 24-72 hrs, 2 and 4 weeks. During each, further DSME was provided, BG logs reviewed, and diabetes medications adjusted as needed by the CDE. Meter and insulin injections skills were reinforced as needed. Outpatient navigation included securing a primary care appointment no later than 4 weeks after study completion. Final contact was via telephone at 90 days. The MMS© (Morisky Medication Adherence Survey) was taken at 2 and 4 weeks and during the final telephone visit. Interim return visits to the ED or admissions to the hospital were queried at each visit. A follow up HbA1C was obtained at week 4 using the POC A1CNow+ ®, and a venous HbA1C was drawn if the POC result was above 13% .
  Other Names: Survival skills self-management education
  Arms: Intervention

SUMMARY:
A 4 week prospective, randomized controlled study was carried out to assess the impact of a care delivery intervention which focused on blood glucose (BG) management among adults with type 2 diabetes presenting to the Emergency Department (ED) with BG > 200mg/dL (11.1 mmol/L). The intervention was designed by a multi-disciplinary team of ED physicians and nurses, endocrinologists and diabetes educators. The intervention incorporated three components: a guideline-based algorithm for diabetes medication management; survival skills diabetes self-management education (DSME); and support for health system navigation. The control group received usual care per the ED's policies and procedures for management of high blood glucose.

DETAILED DESCRIPTION:
We evaluated a concise diabetes care delivery intervention designed to advance glycemic medications and deliver diabetes self-management education (DSME) among adults with type 2 diabetes presenting to the emergency department (ED) with uncontrolled hyperglycemia. The primary hypothesis was that there would be improvement in HbA1c.

A 4 week, randomized controlled trial provided algorithm-based antihyperglycemic medications management, survival skills DSME and navigation to primary care for ED patients with BG > 200mg/dL. Medications were titrated and DSME delivered by endocrinologist-supervised certified diabetes educators. Controls received usual care.

ELIGIBILITY:
Inclusion Criteria:

* A new or existing diagnosis of type 2 diabetes;
* BG > 200 mg/dl in the ED;
* age >/= 18 years;
* willing and able to check BG and self-inject insulin, if required and otherwise stable for discharge to the outpatient setting.

Exclusion Criteria:

* type 1 diabetes and other specific types of diabetes per the American Diabetes Association Position Statement on the Classification of Diabetes Mellitus,
* pregnancy or anticipated conception in the next 3 months;
* treatment with a glucocorticoid, unless at a stable physiologic replacement dose; or
* a history of diabetic ketoacidosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle F Magee, MD, MBBCh, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share IPD. Study results data have been published and shared at national meetings. The PI is open to discussions about the data as requested.

REFERENCES:
- [Background] Magee MF, Nassar C. Hemoglobin A1c testing in an emergency department. J Diabetes Sci Technol. 2011 Nov 1;5(6):1437-43. doi: 10.1177/193229681100500615. PMID 22226261
- [Result] Magee MF, Nassar CM, Copeland J, Fokar A, Sharretts JM, Dubin JS, Smith MS. Synergy to reduce emergency department visits for uncontrolled hyperglycemia. Diabetes Educ. 2013 May-Jun;39(3):354-64. doi: 10.1177/0145721713484593. Epub 2013 Apr 22. PMID 23610182
- [Result] Lewis VR, Benda N, Nassar C, Magee M. Successful patient diabetes education in the emergency department. Diabetes Educ. 2015 Jun;41(3):343-50. doi: 10.1177/0145721715577484. Epub 2015 Mar 24. PMID 25804628

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Diabetes survival skills self-management education (BG meter instruction if the patient did not already have a meter or confirmation of self-BG monitoring technique if they did; instructions on how to self-inject insulin if prescribed; and information on BG targets, signs and treatment of hypoglycemia and hyperglycemia, basic nutrition information and when to call the doctor or go to the ED.); plus diabetes medication management using medication algorithm (Metformin, sulfonylureas and basal insulin were included in the algorithm) by diabetes educator supervised by endocrinologist, plus health system navigation.
  .Diabetes medication management: As above plus- Follow-up intervention visits were at 24-72 hrs, 2 and 4 weeks. During each, further DSME was provided, BG logs reviewed, and diabetes medications adjusted as needed by the CDE. Meter and insulin injections skills were reinforced as needed. Outpatient navigation included securing a primary care
Period: Overall Study
Arm/Group | Intervention | Control
Started | 51 | 50
Completed | 37 | 41
Not Completed | 14 | 9
Not completed — Lost to Follow-up | 14 | 9

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Diabetes survival skills self-management education (G meter instruction if the patient did not already have a meter or confirmation of self-BG monitoring technique if they did; instructions on how to self-inject insulin if prescribed; and information on BG targets, signs and treatment of hypoglycemia and hyperglycemia, basic nutrition information and when to call the doctor or go to the ED. ; plus diabetes medication management using medication algorithm ( Metformin, sulfonylureas and basal insulin were included in the algorithm) by diabetes educator supervised by endocrinologist, plus health system navigation.
  Diabetes medication management: As above plus- Follow-up intervention visits were at 24-72 hrs, 2 and 4 weeks. During each, further DSME was provided, BG logs reviewed, and diabetes medications adjusted as needed by the CDE. Meter and insulin injections skills were reinforced as needed. Outpatient navigation included securing a primary care
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 47 | 95
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (14) | 50 (12) | 50 (13)
Gender [Count of Participants; unit: Participants]
  Female | 31 | 24 | 55
  Male | 20 | 26 | 46
Region of Enrollment [Number; unit: participants]
  United States | 51 | 50 | 101

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1C at 4 Weeks
Description: Hemoglobin A1C at index/baseline visit in the ED and at 4 weeks. A1C was measured using the Bayer A1C-Now+ point of care test system device. If the reading was over 13%, the upper limit of the assay, a venous sample A1C was sent to the hospital lab for analysis.
Time Frame: 4 weeks
Population: Participants who completed the full 4 week study period were included in the primary outcomes analysis.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Intervention | Control
Number analyzed (Participants) | 37 | 41
percentage of glycosylated hemoglobin | 10.5 (1.9) | 11.1 (2.1)

2. Primary Outcome: Medication Adherence
Description: Score on 8 item Modified Morisky Medication Scale used to assess medication adherence. This scale is a structured and widely used self reported questionnaire used to assess medication taking behaviors.The total score ranges from 0 to 8. A score of 0 is considered "high"adherence, 1 to 2 is considered "medium" adherence, and >2 is considered "low" adherence.
Time Frame: 4 weeks
Population: 33 patients in the intervention group and 30 in the control group completed the scale at baseline and at 4 weeks and their data was analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 33 | 30
units on a scale | 1.6 (1.4) | 2.5 (2.2)

3. Secondary Outcome: Blood Glucose < 180mg/dL
Description: Number of patients in each group with BG < 180 mg/dl at 4 weeks from baseline
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 37 | 41
participants | 24 | 11

4. Secondary Outcome: Hypoglycemia
Description: Hypoglycemia was defined as BG < 70mg/dL. Severe hypoglycemia was defined as BG <40mg/dL and/or requiring assistance to treat. We tracked the total number of hypoglycemia episodes in each group.
Time Frame: 4 weeks
Population: we collected data on the total number of hypoglycemia episodes in each group, not the number or participants with hypoglycemia as some participants had more than 1 episode and we wanted to capture those as separate incidents.
Measure: Number; unit: total incidents of hypoglycemia
Arm/Group | Intervention | Control
Number analyzed (Participants) | 37 | 41
total incidents of hypoglycemia | 2 | 1

5. Other Pre Specified Outcome: ED Visits and Hospitalizations
Description: number ED visits and hospitalizations pre and post intervention as self-reported by participants
Time Frame: 12 weeks
Population: Self reported Number of ED visits and hospitalizations 3 months prior to and 3 months after the intervention
Measure: Number; unit: number of ED visits and hospitlizations
Groups:
- Intervention: Diabetes survival skills self-management education; plus diabetes medication management using medication algorithm by diabetes educator supervised by endocrinologist, plus health system naviagation.
  Metformin, sulfonylureas and basal insulin were included in the algorithm. Survival skills DSME included: BG meter instruction if the patient did not already have a meter or confirmation of self-BG monitoring technique if they did; instructions on how to self-inject insulin if prescribed; and information on BG targets, signs and treatment of hypoglycemia and hyperglycemia, basic nutrition information and when to call the doctor or go to the ED.
  Diabetes medication management: As above plus- Follow-up intervention visits were at 24-72 hrs, 2 and 4 weeks. During each, further DSME was provided, BG logs reviewed, and diabetes medications adjusted as needed by the CDE. Meter and insulin injections skills were reinforced as needed. Navigation included securing a primary care
Arm/Group | Intervention | Control
Number analyzed (Participants) | 37 | 41
number of ED visits and hospitlizations | 7 | 10

ADVERSE EVENTS:
Arm/Group | Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/51 | 1/50
Other Adverse Events (participants affected / at risk) | 2/51 | 3/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=51) | Control (N=50)
hospitalization due to exacerbation of gastroperisis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Patient with history of poorly controlled diabetes and of gastroperisis related emergency room visits and hospitlalizations
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=51) | Control (N=50)
hyperglycemia requiring return to Emergency room (Endocrine disorders) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1)
arthritis pain exacerbation (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Not all subjects completed the study, yet dropout rates by arm were similar. Medication adherence was self-reported - concurrent improvement in glycemic control was concordant with its improvement. Impact on ED return visits could not be determined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No